CLINICAL TRIAL: NCT01705561
Title: Evaluation of Attitudes of Premenopausal Latin American Patients With Breast Cancer Towards the Risk of Loss Their Fertility by Chemotherapy
Brief Title: Evaluation of Attitudes About Fertility
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Grupo de Estudios Clínicos Oncológicos Peruano (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: GECOPERU 01-2012
Record Dates: First submitted 2012-10-10; First posted 2012-10-12 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Breast Cancer
Keywords: fertility; chemotherapy; breast cancer; latin american women; pre menopausal
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
* Assess the attitudes and feelings of premenopausal Latin American women towards the risk of loss their fertility by adjuvant chemotherapy.
* Correlate the attitudes with other variables including age at diagnosis, already having children, number of children, level of instruction, marital status, frequency of menstrual cycle.

DETAILED DESCRIPTION:
Eligibility criteria:

* Latin American women with evidence of cancer diagnosis at premenopausal status
* Over 18 years
* Agree to sign the informed consent
* No evidence of infertility.

ELIGIBILITY:
Inclusion Criteria:

* women with breast cancer diagnosis in premenopausal
* over 18 years
* signed informed consent

Exclusion Criteria:

* Evidence of infertility at diagnosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women with diagnosis of breast cancer in pre menopausal status
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2012-12; Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: HENRY L GOMEZ, DR, Principal Investigator — Grupo de Estudios Clínicos Oncológicos Peruano
Locations (2):
- Peru (2):
  - Instituto Nacional de Enfermedades Neoplasicas, Lima, Lima Province
  - Oncosalud, Lima, Lima Province